CLINICAL TRIAL: NCT06830369
Title: Effect of a Virtual Reality Program on Patient Comfort in the Surgical Intensive Care Unit of a French University Hospital: Study Protocol for a Monocentric, Prospective, Superiority, Randomized Controlled Trial, With Blinded End-point (PROBE), ZION Study
Brief Title: Effect of a Virtual Reality Program on Patient Comfort in the Surgical Intensive Care Unit
Acronym: ZION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PI2024_843_0082
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Immersive Virtual Reality; Discomfort; IPREA; Intensive Care Unit; Delirium
Keywords: Immersive virtual reality; discomfort; IPREA; intensive care unit; delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (Active Comparator)
  Interventions: Other: usual health care
- intervention group (Experimental)
  Interventions: Device: HypnoVR

INTERVENTIONS:
Device: HypnoVR — In the intervention group, after extubation, patients will receive IVR with HypnoVR®, twice-a-day over two to five days. The product consists of HypnoVR® virtual reality software and HypnoVR® Compagnon remote control software. HypnoVR® is a CE-marked class 1 medical device, developed and marketed by HypnoVR SAS, an ISO 13484:2016 and ISO 27001:2017 certified company. The device works with a virtual reality headset, a personal audio device and a mobile terminal. The investigators will only use sessions of 10 to 20 minutes. For each type of session, a visual universe, a musical atmosphere and a male or female voice are defined. Typically, the scenarios include 3 phases: preparation, hypnosis and return. We will use the following sessions: anxiety, pain, rehabilitation.
  Arms: intervention group
Other: usual health care — usual health care
  Arms: standard group

SUMMARY:
Admission to a surgical intensive care unit (ICU) following major surgery is associated with a number of discomforts, not only related to the disease itself, but also to the care provided or the ICU environment itself (lights, sounds, pain, sleep deprivation, thirst...). This discomfort is real, and can be associated with psychological consequences. The investigators hypothesized that the use of immersive virtual reality (IVR) with HypnoVR® is feasible and can help reduce discomfort in intensive care.The ZION trial is a prospective, monocentric trial, randomizing 194 patients admitted in a surgical intensive care unit after a major surgery. The inclusion criterion are patients admitted in a surgical intensive care for at least 48 hours following major surgery (cardiac, thoracic or major abdominal surgery). Patients will be allocated to the intervention group (n=97) or the control group (n=97). In the intervention group, patients will receive IVR using HypnoVR®, twice a day, during the ICU stay (2 to 5 days). In the control group, postoperative care will be conducted according to standard cares without IVR. The primary endpoint will be the 18-items IPREA questionnaire on the day of ICU discharge. The secondary endpoints will include intensity of discomfort symptoms (anxiety, pain, dyspnea, thirst and sleep deprivation), incidence of delirium, cumulative morphine consumption at ICU discharge, length of ICU stay, and anxiety or depression at 1 month after discharge from intensive care and patient experience of device use.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* scheduled for a major surgery (cardiothoracic surgery or a major abdominal surgery)
* Written informed consent from patient.
* Admitted in a surgical ICU for a postoperative care for at least 48 hours.
* Absence of delirium at inclusion (RASS and CAM-ICU scale)

Exclusion Criteria:

* Missing informed consent
* Patient strictly under 18 years old
* Inclusion in other study within the last 30 days
* Pregnancy
* Emergency hospitalization
* Progressive sepsis
* Patient transferred from another intensive care unit
* Short-term life-threatening condition
* Active psychiatric illness requiring antidepressant, antipsychotic or anxiolytic treatment
* Mechanical ventilation > 48 hours
* Patient known to have cognitive disorders.
* Unbalanced epilepsy
* Visual problems (absence of binocular vision, blindness) and/or auditory problems (deafness) preventing the use of virtual reality
* Pregnant or breast-feeding women
* Patients under guardianship or deprived of their liberty
* Patients not registered with the national social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
IPREA questionnaire value | at the day of ICU-discharge from intensive care, within 5 days
  The primary endpoint will be the 18-item IPREA questionnaire on the day of ICU discharge from intensive care. Each item of the questionnaire includes factors such as noise, light, bed, sleep, thirst, hunger, cold, heat, pain, medical device, intimacy, anxiety, isolation, visiting hours, phone, information, breath and depression. It represents a valid French questionnaire on self-perceived discomfort in intensive care, which is the only discomfort assessment instrument validated for use in the ICU.

SECONDARY OUTCOMES:
Intensity of discomfort symptoms | at the day of ICU-discharge from intensive care, within 5 days
  The intensity of the following discomfort symptoms assessed on the day of discharge from intensive care (within 5 days) : anxiety, pain, dyspnea, thirst and sleep deprivation. The intensity of these discomforts will be assessed using a NRS ranging from 0 to 10 (0 = no discomfort; 10 = worst possible symptom).
Delirium incidence | daily until ICU discharge (within 5 days)
  The incidence of delirium measured using the CAM-ICU and RASS scale, daily until discharge from intensive care.
  RASS is the Richmond agitation & sedation scale (RASS) The RASS score ranges from a score of -5, where a patient is deemed "unarousable", to a score of +4, where a patient is "violent and immediate danger to staff". If the RASS score is too low (less than -3), meaning that the patient is too drowsy or sedated, then the CAM-ICU cannot be performed .
  CAM-ICU is : The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) is a tool specifically designed to assess for delirium in the context of ICU patients, including those on mechanical ventilation.
  The final CAM-ICU- score is positive for delirium or negative for delirium.
Cumulative opioid consumption (morphine or oxycodone) | At ICU discharge day (within 5 days)
  Cumulative opioid consumption (morphine or oxycodone) expressed in milligrams at discharge from intensive care,
Length of stay (in days) | At ICU discharge day (within 5 days)
  Length of stay is defined in days between admission to intensive care and discharge from the hospital.
Anxiety and depression at 1 month | at 1 month after discharge from intensive care
  Anxiety and depression at 1 month (V2 follow-up visit) after discharge from intensive care using the HAD scale.
  HAD scale is : Hospital Anxiety and Depression Scale (HADS) is a 14-item scale, with seven items relating to anxiety and seven relating to depression.
  Scores are :
  0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Patient experience score | At ICU discharge day (within 5 days)
  Patient experience of device use on discharge from intensive care, using a numeric scale from 1 to 5.
  1. Dissatisfied / did not wish to repeat the experience
  2. Not very satisfied with the experience
  3. Moderately satisfied with the experience
  4. Satisfied with the experience
  5. Very satisfied / Would like to repeat the experience

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huette P, Malaquin S, Lefebvre T, Devos C, Ibrahima A, Daumin C, Coupez A, Josse E, Besserve P, Haye G, Bayart G, Guilbart M, Gibert L, Beyls C, Dupont H, Meynier J, Diouf M, Mahjoub Y, Abou-Arab O. Effect of a virtual reality program on patient comfort in the surgical intensive care unit of a French university hospital: study protocol for a monocentric, prospective, superiority, randomised controlled trial-ZION study. BMJ Open. 2025 Jul 17;15(7):e101243. doi: 10.1136/bmjopen-2025-101243. PMID 40675645